CLINICAL TRIAL: NCT05904457
Title: A Phase II Clinical Trial of Bevacizumab Plus eRlotinIb in patientS With Advanced Cancer Having Genetic Alterations in Krebs Cycle (BRISK, KCSG AL22-16)
Brief Title: A Phase II Stydy of Bevacizumab Plus Erlotinib in Patients for Krebs Cycle Altered Cancer
Acronym: BRISK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Inkeun Park, Clinical Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCT0007840
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumors; Advanced Solid Tumors; Metastatic Cancer
Keywords: Krebs cycle; FH; IDH; SDH; bevacizumab; erlotinib; cancer; aerobic glycolysis; brisk
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: erlotinib

INTERVENTIONS:
Drug: bevacizumab — Patients will receive bevacizumab 10 mg/kg IV over 30-90 minutes every 2 weeks until disease progression or unacceptable toxicity.
  Other Names: onbevzi
Drug: erlotinib — Patients will receive elrotinib 150 mg orally once a day continuously until disease progression or unacceptable toxicity.
  Other Names: eltinib

SUMMARY:
A national, prospective, multi-center, open-label, single arm phase II trial investigating the efficacy and safety of bevacizumab plus erlotinib in patients with advanced cancers which harbors genomic alterations in Krebs cycle

DETAILED DESCRIPTION:
The BRISK study will recruit patients with locally advanced or metastatic solid tumor harboring the genomic alterations in Krebs cycle (e.g. fumarate hydratase, isocitrate dehydrogenase, succinate dehydrogenase) who had disease progression on standard systemic treatment and/or has no standard treatment option, and investigate the efficacy and safety of bevacizumab plus erlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the KOSMOS-II master trial
2. Age 19 or more
3. Histologically confirmed solid cancer
4. Genetic alteration in genes related to Krebs cycle (fumarate hydratase, succinate dehydrogenase, isocitrate dehydrogenase, or maleate dehydrogenase 2). Only pathogenic and likely pathogenic variant in either germline or somatic gene will be permitted.
5. Patients with locally advanced, recurrent, or metastatic disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
6. Disease progressed during or after standard treatment with no further treatment option, no standard treatment, patient's refusal to receive standard treatment, or unfit for standard treatment. If standard treatment contains bevacizumab and/or erlotinib, patient can be included according to treating physician's discretion
7. Measurable disease according to RECIST v1.1 criteria
8. ECOG performance status 0 or 2
9. Adequate bone marrow, hepatic, and renal function Hematology

   * Neutrophil >= 1,500/mm3
   * Platelet >= 100,000/mm3
   * Hemoglobin >= 9 g/dL Liver function tests
   * Total bilirubin ≤ 1.5 xULN
   * AST, ALT ≤ 3 xULN (in case of liver metastasis, 5 x upper limit of normal) Renal function tests
   * Creatinine clearance >= 30 mL/min
10. Life expectancy more than 3 months
11. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Previous treatment with combination of vascular endothelial growth factor inhibitors and epithelial growth factor receptor inhibitors. Previous exposure to only VEGF inhibitor or EGFR inhibitor, or sequential exposure to both agents can be included at the treating physician's discretion
2. Previous radiotherapy to the only measurable lesion: but previous radiotherapy will be permitted unless the lesion is the only measurable lesion
3. Uncontrolled CNS metastasis (brain and/or leptomeningeal metastasis) that requires anti-edema drugs such as steroid for symptoms or symptom management. Primary CNS malignancy such as glioblastoma can be included by treating physician's discretion.
4. Have clinically problematic cardiovascular diseases, such as unstable angina, congestive heart failure, advanced arrhythmia requiring treatment with medication, or a history of myocardial infarction within 12 months prior to enrollment. Inclusion is allowed if patient has no evidence of active disease for at least 6 months prior to enrollment.
5. Inadequately controlled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications).
6. History of cerebral vascular accident (CVA) or transient ischemic attack (TIA) ≤ 6 months prior to screening
7. History of bleeding diathesis or coagulopathy
8. Urine dipstick proteinuria≥2+ or urine protein/creatinine ratio >1.0. If patients are discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of proteinuria in 24 hours.
9. Currently on maximal dose of therapeutic anticoagulation for thromboembolic disease.
10. Clinically significant bleeding (hemoptysis, melena, hematochezia, tumor bleeding, etc.), or at risk of significant bleeding (tumor infiltrating into the great vessels or an evident cavitation of cancer lesions)
11. Have any of the following gastrointestinal disturbances.

    * Unable to take internal medications ② Required intravenous feeding ③ Have malabsorption due to surgical treatment (such as gastrointestinal resection) or underlying disease ④ Have an active peptic ulcer (enrollment is permitted if the patient is being given prophylactic treatment for a previous condition or treatment for complications from gastritis, etc.) ⑤ History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess ≤ 6 months prior to screening
12. Serious non-healing wound, ulcer, bone fracture or have undergone a major surgical procedure, open biopsy, or significant traumatic injury ≤28 days prior to screening.
13. Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri or prostate cancer and curatively treated thyroid cancer of any stage.
14. Pregnancy or breast feeding
15. Men or women who are not intending to use contraceptive methods during the study period.
16. Major surgery is scheduled during the study period
17. Other severe acute or chronic medical or psychiatric condition
18. Individuals who are deemed to be unsuitable for participation in this study by the investigators for any other reason
19. Where participation in this clinical trial is not appropriate in the judgment of the investigator for any other reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months after treatment initiation (estimated average)
  Defined as a proportion of complete response (CR) + partial response (PR) according to RECIST v1.1, the fraction with a response (CR+PR) will be reported separately by cohort, along with a 95% confidence interval

SECONDARY OUTCOMES:
Progression-free survival | Time from study treatment initiation until disease progression or death, assessed up to 1 years from study enrollment (estimated average)12 months after treatment initiation (estimated average)
  Assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, PFS will be determined using the Kaplan-Meier method, and the curves presented along with a 95% confidence interval on the median PFS
Overall survival (OS) | Time from study treatment initiation until death from any cause, assessed up to 2 years from study enrollment (estimated average)
  The Kaplan-Meier method will be used and the curves presented along with a 95% confidence interval on the median OS
Incidence of adverse events | Time from study treatment initiation up to 30 days after last treatment, 12 months after treatment initiation (estimated average)
  Severity of adverse events will be graded by NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events) v5.0

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Cha University Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Yonsei Cancer Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan